CLINICAL TRIAL: NCT05476497
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of VLP Peanut in Healthy Subjects and Subjects With Peanut Allergy and to Explore Preliminary Signals of Its Efficacy (PROTECT)
Brief Title: Phase I Trial to Evaluate VLP Peanut in Healthy and Peanut Allergic Subjects
Acronym: PROTECT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VLP-Peanut101
Record Dates: First submitted 2022-07-08; First posted 2022-07-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Two part clinical trial:
  Part A- Open-label with two groups (A1 and A2):
  i) A1 (Healthy Subjects): subcutaneous (SC) dosing with ascending concentrations of VLP Peanut.
  ii) A2 (peanut allergic subjects): skin prick test (SPT) performed with ascending concentrations of VLP Peanut.
  Part B - double-blind, placebo-controlled part that will enroll Peanut Allergic Subjects: subcutaneous (SC) dosing with ascending concentrations of VLP Peanut.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A is open label. Part B is double blind, placebo controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Group A1 (Experimental): 4 parallel cohorts (1-4) of adult healthy subjects. Each cohort will receive 6 ascending subcutaneous administrations of VLP Peanut.
  Interventions: Biological: VLP Peanut
- Part A - Group A2 (Experimental): Adult peanut allergic subjects, will undergo skin prick tests with ascending concentrations of VLP Peanut.
  Interventions: Biological: VLP Peanut
- Part B - Cohorts 1-4 (Experimental): 4 parallel cohorts (1-4) of peanut allergic subjects. Each cohort will receive 6 ascending subcutaneous administrations of VLP Peanut.
  Interventions: Biological: VLP Peanut; Biological: Placebo

INTERVENTIONS:
Biological: VLP Peanut — solution for subcutaneous administration
  Arms: Part A - Group A1; Part B - Cohorts 1-4
Biological: Placebo — solution for subcutaneous administration
  Arms: Part B - Cohorts 1-4
Biological: VLP Peanut — solution for Skin-prick testing
  Arms: Part A - Group A2

SUMMARY:
This phase I clinical trial is designed to evaluate the safety and tolerability of VLP Peanut in healthy subjects and in subjects with peanut allergy (PA). This clinical trial will evaluate the immunotoxicity profile of VLP Peanut in healthy subjects and assess the immunotoxicity profile and the degree of reactogenicity (allergenicity) in subjects with PA. This clinical trial will also explore preliminary proof of efficacy of VLP Peanut in subjects with PA.

ELIGIBILITY:
Part A Main Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Subject who has a signed and dated Informed Consent Form (ICF).
3. Subject must be 18 to 50 years inclusive, at the time of signing the ICF.
4. Male or female.
5. Female subjects who are not of childbearing potential (or females of childbearing potential who agree to comply with the contraceptive requirements of the clinical trial protocol).
6. Good general health, as determined by the Investigator.
7. A positive SPT to histamine.

   The following additional inclusion criteria are only applicable to the healthy subjects in Group A1:
8. Healthy subjects (non-atopic) with no clinically significant co-morbidity (including broncho-reactive airway disease like asthma, current allergic rhinitis, etc.).
9. Subjects with no history of allergy or intolerance to peanut or any other food and who consume peanuts with no effect.
10. Subjects with lack of sensitivity to peanut allergen confirmed by SPT using whole peanut extract.
11. Peanut specific immunoglobulin E (IgE) <0.35 kU/L.
12. Ara h 2 specific IgE <0.35 kU/L.
13. Subjects with negative basophil activation test (BAT).

    The following additional inclusion criteria are only applicable to the subjects with PA in Group A2:
14. Clinical history of physician diagnosed PA.
15. Peanut allergen sensitivity confirmed by SPT and IgE.
16. Subjects who currently adhere to a strict peanut-free diet and who agree to continue this for the duration of the clinical trial.
17. Subjects who are able to handle and correctly use an adrenaline auto-injector.

Part B Main Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Subject who has a signed and dated ICF.
3. Subjects aged 18 to 50 years of age inclusive, at the time of signing the ICF.
4. Male or female.
5. Female subjects who are not of childbearing potential (or females of childbearing potential who agree to comply with the contraceptive requirements of the clinical trial protocol).
6. Clinical history of physician diagnosed PA.
7. Peanut allergen sensitivity confirmed by positive SPT and Ara h 2 specific IgE ≥1.0 kU/L
8. Subjects with positive BAT.
9. Subjects who currently adhere to a strict peanut-free diet and who agree to continue this for the duration of the clinical trial.
10. Good general health, as determined by the Investigator.
11. Subjects who are able to handle and correctly use an adrenaline auto-injector.

Main Exclusion Criteria Part A and B:

1. Pregnant or lactating subject.
2. Presence of any medical condition that may reduce the ability to survive a serious allergic reaction.
3. Subjects with atopic dermatitis with >25% skin surface involvement.
4. For subjects with PA, presence of severe, poorly controlled or uncontrolled asthma.
5. History of severe or life-threatening anaphylactic reactions to peanut resulting in neurological compromise or requiring mechanical ventilation.
6. History of severe or life-threatening anaphylactic reactions to foods (excluding peanuts), insect venom, exercise, drugs, or idiopathic causes, resulting in neurological compromise or requiring mechanical ventilation or deemed severe as per Investigator assessment.
7. Unable to receive epinephrine therapy or at greater risk of developing adverse reactions after epinephrine administration as assessed by the site Investigator.
8. Clinical history of drug or alcohol abuse, which, in the Investigator's opinion, could interfere with the subject's ability to participate in the clinical trial.
9. Participation in a clinical research trial with any investigational drug/placebo within 3 months of screening (Visit 1) or concomitantly with this clinical trial.
10. Personal, financial or other dependent relationship (e.g., employee or immediate relative) with the clinical trial site, Sponsor, Sponsor's representative, or another individual who has access to the clinical trial protocol.
11. Vulnerable subjects or those in judicial or governmental detention, detainment or imprisonment in a public institution.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number and severity of Adverse Events (AEs) (including local and systemic AEs). | Group A1: 18 weeks; Part B: 64 weeks (Part B). Group A2: 3 days.
Number of subjects discontinuing prematurely from treatment due to AEs | Group A1: 11 weeks Part B: 15 weeks

SECONDARY OUTCOMES:
Incidence of fatigue (tiredness) | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of fatigue (tiredness) | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of headache | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of headache | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of muscle pain | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of muscle pain | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of cough | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of cough | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of sore throat | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of sore throat | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of runny nose | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of runny nose | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of chills | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of chills | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Incidence of fever (i.e. body temperature equal or above 38ºC (100.4ºF)) | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Frequency of fever (i.e. body temperature equal or above 38ºC (100.4ºF)) | Group A1: 14 weeks Part B: 16 weeks
  Part of solicited pre-specified influenza like symptoms in healthy and peanut allergic subjects.
Wheal sizes after SPT in subjects with PA (Part A only) | 15-20 minutes after skin pricking
  wheal diameter (longest diameter)
Respiratory and Cardiovascular System Alterations as assessed by brief physical examination | On each dosing day - Group A1/Group part B: pre-dose and 30+/-10 minutes post dose; Group A2: pre-skin pricking and 1 hour post-skin pricking
  Assessment of the respiratory and cardiovascular systems through palpation, auscultation and percussion that are performed by physician to identify any potential abnormalities
Alterations in the lung function | Group A1 and Group Part B: On each dosing day pre-dose and 30 to 60 minutes post-dose; Group A2: pre skin pricking and 1 hour post skin pricking
  Spirometry test. Alteration is considered when values obtained are: Forced expiratory volume in one second (FEV1) <80% of predicted with a FEV1/Forced vital capacity (FVC) ratio <75%.
Alterations in urine pH | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Urinalysis Dip-stick: pH
Alterations in urinalysis (protein) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: protein
Alterations in urinalysis (glucose) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: glucose
Alterations in urinalysis (ketones) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: ketones
Alterations in urinalysis (urobilinogen) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: urobilinogen
Alterations in urinalysis (bilirubin) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: bilirubin
Alterations in urinalysis (nitrite) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: nitrite
Alterations in Urinalysis (blood) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: blood
Alterations in Urinalysis (leukocytes) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Dip-stick: leukocytes
Alterations in Serum Chemistry (Glucose) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: Glucose
Alterations in Serum Chemistry (Sodium) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: sodium
Alterations in Serum Chemistry (Uric Acid) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: uric acid
Alterations in Serum Chemistry (Urea) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: urea
Alterations in Serum Chemistry (potassium) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: potassium.
Alterations in Serum Chemistry (Calcium) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: calcium.
Alterations in Serum Chemistry (Creatinine) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: creatinine.
Alterations in Serum Chemistry (chloride) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: chloride
Alterations in Serum Chemistry (total protein) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: total protein
Alterations in Serum Chemistry (phosphorus) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: phosphorus
Alterations in Serum Chemistry (cholesterol) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: cholesterol
Alterations in Serum Chemistry (albumin) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: albumin
Alterations in Serum Chemistry (total bilirubin) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: total bilirubin
Alterations in Serum Chemistry (alkaline phosphatase) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: alkaline phosphatase
Alterations in Serum Chemistry (lactate dehydrogenase) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: lactate dehydrogenase (LDH)
Alterations in Serum Chemistry (aspartate aminotransferase) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: aspartate aminotransferase (AST).
Alterations in Serum Chemistry (Alanine aminotransferase) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: Alanine aminotransferase (ALT)
Alterations in Serum Chemistry (gamma-glutamyl transferase) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: gamma-glutamyl transferase (GGT)
Alterations in Serum Chemistry (C-reactive protein) | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Detection of the levels of: C-reactive protein (CRP).
Alterations in hemoglobin levels | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Hematology, analysis Hemoglobin levels
Alterations in the hematocrit | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Hematology, analysis of the hematocrit
Alterations in Red Blood Cells (RBC) levels | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Hematology, analysis of total RBC and RBC indices
Alterations in White Blood Cells (WBC) levels | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Hematology: total WBC and differentials
Platelet counts alterations | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  Hematology: platelet count
Serum/Urine Pregnancy Test | Group A1: 18 weeks; Group A2: 2-5 days; Part B: 16 weeks
  In all females of childbearing potential. Serum test at V1 and Urine test at subsequent visits. Confirmatory serum pregnancy test to be conducted if urine test is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter-Jan De Kam, PhD, Study Director — Allergy Therapeutics
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Trio Clinical Trials, LLC., Houston, Texas
  - University of Wisconsin School of Medicine and Public Health Asthma, Allergy, and Pulmonary Clinical Research, Madison, Wisconsin

REFERENCES:
- [Derived] Layhadi JA, Starchenka S, De Kam PJ, Palmer E, Patel N, Keane ST, Hikmawati P, Drazdauskaite G, Wu LYD, Filipaviciute P, Parkin RV, Oluwayi K, Rusyn O, Skinner MA, Heath MD, Hewings SJ, Kramer MF, Turner P, Shamji MH. Ara h 2-expressing cucumber mosaic virus-like particle (VLP Peanut) induces in vitro tolerogenic cellular responses in peanut-allergic individuals. J Allergy Clin Immunol. 2025 Jan;155(1):153-165. doi: 10.1016/j.jaci.2024.08.010. PMID 39756833